CLINICAL TRIAL: NCT03387735
Title: Heart-Related Multiple Chronic Conditions in Primary Care: Behavioral Technology
Brief Title: Multiple Chronic Conditions for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Medical University of South Carolina (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2017-0849; A195010 (Other: UW Madison); ENGR\INDUSTRIAL ENGR\CHESS (Other: UW Madison); 1R01HL134146-01A1 (NIH)
Record Dates: First submitted 2017-11-02; First posted 2018-01-02 (Actual); Results first posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Chronic Disease
Keywords: Hypertension, Hyperlipidemia, Diabetes, Arthritis, Obesity
MeSH Terms: conditions — Chronic Disease; Hypertension; Hyperlipidemias; Diabetes Mellitus; Arthritis; Obesity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) + Internet (Placebo Comparator): Patients will be given access to helpful websites such as National Institute on Aging.
  Interventions: Other: Treatment as usual (TAU) + Internet
- Treatment as usual (TAU) + ElderTree (Experimental): Patients will be given access to the ElderTree website for 12 months which provides tools, motivation, and social support to help them manage their specific set of chronic conditions and communicate with peers and their primary care physician.
  Interventions: Behavioral: TAU + ElderTree

INTERVENTIONS:
Other: Treatment as usual (TAU) + Internet — Patients in this group will receive TAU+internet and links to helpful websites.
  Arms: Treatment as usual (TAU) + Internet
Behavioral: TAU + ElderTree — For the patient, ElderTree provides tools, motivation, and social support to help them manage their specific set of chronic conditions and communicate with peers and their primary care physician.
  For the clinic, ElderTree has a Clinician Report (CR), a visual dashboard of health-tracking data that can be customized based on the needs of the clinic. The CR provides alerts to the clinician when a patient passes a certain threshold. The dashboard is intended to help clinicians prepare for patient office visits.
  Arms: Treatment as usual (TAU) + ElderTree

SUMMARY:
Multiple chronic conditions are common and expensive among patients aged ≥65 and are associated with lower quality of life, poorer response to treatment, worse medical and psychiatric outcomes, higher mortality, and higher costs of care.

The primary purpose of this study is to conduct a randomized clinical trial (RCT) to examine the effects of ElderTree --a web-based intervention--on health outcomes and healthcare use among older adults with several chronic health conditions, such as diabetes, high blood pressure, high cholesterol, COPD, BMI over 30, congestive heart failure, chronic kidney disease, arrhythmia/atrial fibrillation, chronic pain, arthritis.

The investigator's hypothesis is that patients assigned to TAU+ElderTree will have better quality of life and fewer primary care visits than those assigned to TAU+Internet.

ELIGIBILITY:
Inclusion Criteria:

1. are ≥65 years old
2. have been treated in the University of Wisconsin Health clinics for at least the previous 18 months with no plans to leave during the study period
3. have 3 or more of the following chronic conditions: hypertension, hyperlipidemia, diabetes, arthritis, BMI over 30, chronic kidney disease, congestive heart failure, arrhythmia/atrial fibrillation, pulmonary heart disease or pulmonary vascular disease, chronic pain, COPD
4. report no current psychotic disorder that would prevent participation
5. have no acute medical problem requiring immediate hospitalization
6. be able to read and sign the consent form in English
7. have no known terminal illness
8. be willing to share health-related study data and

   * Systolic and diastolic BP
   * Weight
   * BMI
   * HDL/LDL
   * HbA1C
   * pain score
   * lung function
   * health care utilization: number of ER visits, urgent care visits, primary care visits and specialty care visits
9. allow researchers to share information with their primary care physician

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 346 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Gustafson, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Health Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gustafson DH Sr, Mares ML, Johnston D, Vjorn OJ, Curtin JJ, Landucci G, Pe-Romashko K, Gustafson DH Jr, Shah DV. An eHealth Intervention to Improve Quality of Life, Socioemotional, and Health-Related Measures Among Older Adults With Multiple Chronic Conditions: Randomized Controlled Trial. JMIR Aging. 2024 Dec 6;7:e59588. doi: 10.2196/59588. PMID 39642938
- [Derived] Gustafson DH Sr, Mares ML, Johnston DC, Mahoney JE, Brown RT, Landucci G, Pe-Romashko K, Cody OJ, Gustafson DH Jr, Shah DV. A Web-Based eHealth Intervention to Improve the Quality of Life of Older Adults With Multiple Chronic Conditions: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Feb 19;10(2):e25175. doi: 10.2196/25175. PMID 33605887

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted from January 2018 to December 2019. The intervention period ended in June 2021.
Pre-assignment Details: Two participants signed the consent form and were randomized but did not start the study. One couldn't use the ET website due to macular degeneration. The other one decided he's not interested in using computers and ElderTree.
Groups:
- Treatment as Usual (TAU) + ElderTree: Patients will be given access to the ElderTree website for 12 months which provides tools, motivation, and social support to help them manage their specific set of chronic conditions and communicate with peers and their primary care physician.
  TAU + ElderTree: For the patient, ElderTree provides tools, motivation, and social support to help them manage their specific set of chronic conditions and communicate with peers and their primary care physician.
  For the clinic, ElderTree has a Clinician Report (CR), a visual dashboard of health-tracking data that can be customized based on the needs of the clinic. The CR provides alerts to the clinician when a patient passes a certain threshold. The dashboard is intended to help clinicians prepare for patient office visits.
Period: Overall Study
Arm/Group | Treatment as Usual (TAU) + Internet | Treatment as Usual (TAU) + ElderTree
Started | 168 | 176
Completed | 160 | 160
Not Completed | 8 | 16
Not completed — Lost to Follow-up | 4 | 8
Not completed — Death | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual (TAU) + Internet | Treatment as Usual (TAU) + ElderTree | Total
Number analyzed (Participants) | 168 | 176 | 344
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.54 (6.45) | 75.03 (6.27) | 74.79 (6.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 106 | 209
  Male | 65 | 70 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 167 | 176 | 343
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 8 | 22
  White | 153 | 164 | 317
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 168 | 176 | 344
Health Insurance type [Count of Participants; unit: Participants]
  Medicare | 57 | 69 | 126
  Medicaid | 2 | 1 | 3
  Affordable Care Act | 0 | 0 | 0
  Military | 0 | 0 | 0
  Private insurance | 3 | 2 | 5
  Covered under someone else | 0 | 0 | 0
  No insurance | 0 | 0 | 0
  NA | 1 | 1 | 2
  More than one source | 105 | 103 | 208

OUTCOME MEASURES:

1. Primary Outcome: PROMIS Global Health Measure Score
Description: Quality of life is assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health measure. For consistency with other measures, the time frame has been modified to refer to the past 2 weeks. Scores are calculated using the HealthMeasures Scoring Service. Scores are a T-score metric with a mean of 50 and a standard deviation of 10 with a range of about 20 to 80. Higher scores indicate better quality of life.
Time Frame: Measured at baseline and 12 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Treatment as Usual (TAU) + Internet | Treatment as Usual (TAU) + ElderTree
Number analyzed (Participants) | 168 | 176
T-score
  Baseline: Mental | 46.27 (7.42) | 46.21 (7.16)
  12 Months: Mental | 44.92 (6.82) | 46.38 (7.34)
  Baseline: Physical | 42.40 (6.50) | 42.35 (5.99)
  12 Months: Physical | 42.13 (6.30) | 42.41 (6.32)

2. Primary Outcome: Psychological Flourishing Scale
Description: Psychological well-being is assessed using the Psychological Flourishing Scale. The wording of items has been somewhat modified, including simplifying double-barreled items. For example, "I lead a purposeful and meaningful life" is shortened to "I lead a meaningful life." Scores are a sum of all items with a range from 8 to 40. Higher scores indicate a better well-being.
Time Frame: Baseline and 12-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual (TAU) + Internet | Treatment as Usual (TAU) + ElderTree
Number analyzed (Participants) | 168 | 176
score on a scale
  Baseline | 31.55 (5.39) | 31.12 (5.08)
  12-months | 31.50 (5.15) | 31.48 (5.60)

3. Primary Outcome: UCLA Loneliness Scale
Description: Loneliness is measured using the 8 items from the UCLA Loneliness Scale with the highest factor loadings among older adults. Scores ranged from 8 to 40. Higher scores indicate more loneliness.
Time Frame: Baseline and 12-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual (TAU) + Internet | Treatment as Usual (TAU) + ElderTree
Number analyzed (Participants) | 168 | 176
score on a scale
  Baseline | 16.02 (5.77) | 17.12 (6.04)
  12-months | 16.05 (6.27) | 16.75 (5.86)

4. Secondary Outcome: Unhealthy Laboratory Scores
Description: Laboratory scores are obtained from the patient's electronic health record (EHR) including blood pressure, HAC1 for diabetes, cholesterol, BMI. Some participants did not have this data. The final score is a fraction of the number of unhealthy labs over each persons total labs. Scores range from 0 to 1. Higher scores indicate more unhealthy lab records.
Time Frame: 12-months
Measure: Mean (Standard Deviation); unit: fraction of unhealthy lab scores
Arm/Group | Treatment as Usual (TAU) + Internet | Treatment as Usual (TAU) + ElderTree
Number analyzed (Participants) | 131 | 131
fraction of unhealthy lab scores | 0.64 (0.31) | 0.64 (0.34)

5. Secondary Outcome: Falls
Description: Falls were assessed by asking how often the participant had fallen in the past 3 months. A fall is defined in the survey as "the body going to the ground without being pushed." Here we report statistics for how many times participants had fallen. Falls ranged from 0 to 14.
Time Frame: Baseline and 12-months
Measure: Mean (Standard Deviation); unit: falls
Arm/Group | Treatment as Usual (TAU) + Internet | Treatment as Usual (TAU) + ElderTree
Number analyzed (Participants) | 168 | 176
falls
  Baseline | 0.36 (0.95) | 0.36 (0.88)
  12-months | 0.36 (0.89) | 0.72 (4.09)

6. Secondary Outcome: Symptom Distress
Description: Symptom distress is assessed using a combined list of 20 symptoms and chronic conditions from the General Symptom Distress Scale and Bayliss Disease Burden Scale, assessing the severity of distress for each over the past 2 weeks (0=do not have this, 1=not very distressing, and 5=extremely distressing). Scores range from 0 to 100. Higher scores indicate more symptom distress.
Time Frame: Baseline and 12-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual (TAU) + Internet | Treatment as Usual (TAU) + ElderTree
Number analyzed (Participants) | 168 | 176
score on a scale
  Baseline | 21.10 (14.56) | 20.58 (14.55)
  12-months | 18.86 (14.89) | 18.58 (14.14)

7. Secondary Outcome: Medication Adherence
Description: Medication adherence is assessed with 8 items, 6 based on the Brief Medication Questionnaire by Svarstad et al. We simplified response options so that participants rate how often they had specific issues with medication (1=never and 5=always). On the basis of patients' experiences, we added 2 original items, "Feels like I no longer need it" and "Feels like I don't need the full dose. There were 8 items in total, summed to get a final score. Scores ranged from 8 to 40. Higher scores indicate less medication adherence.
Time Frame: Baseline and 12-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual (TAU) + Internet | Treatment as Usual (TAU) + ElderTree
Number analyzed (Participants) | 168 | 176
score on a scale
  Baseline | 13.14 (4.36) | 13.07 (3.88)
  12-months | 12.70 (4.23) | 12.56 (4.07)

8. Secondary Outcome: Crisis Health Care Visits
Description: Crisis health care was the total number of urgent care visits, emergency room visits, and hospitalizations combined. Reported is the average count of visits. Higher numbers indicate more visits.
Time Frame: Baseline and 12-months
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Treatment as Usual (TAU) + Internet | Treatment as Usual (TAU) + ElderTree
Number analyzed (Participants) | 168 | 176
visits
  Baseline | 0.42 (0.90) | 0.45 (1.06)
  12-months | 0.86 (1.76) | 0.76 (1.45)

9. Secondary Outcome: Long-term Care
Description: Long-term care was the number of nights spent in assisted living facilities and nursing homes over the past 3 months. Number of nights ranged from 0 to 92. Higher numbers indicate more nights spent.
Time Frame: Baseline and 12-months
Measure: Mean (Standard Deviation); unit: nights
Arm/Group | Treatment as Usual (TAU) + Internet | Treatment as Usual (TAU) + ElderTree
Number analyzed (Participants) | 168 | 176
nights
  Baseline | 0.01 (0.15) | 0.25 (2.50)
  12-months | 0.79 (7.76) | 0.29 (2.11)

10. Secondary Outcome: Falls Requiring Medical Attention
Description: Falls requiring medical attention was assessed by one item counting the number of times in the past 3 months. A fall is defined in the survey as "the body going to the ground without being pushed." Here we report statistics for how many times participants had fallen and required medical attention. Falls needing medical attention ranged from 0 to 4.
Time Frame: Baseline and 12-months
Measure: Mean (Standard Deviation); unit: falls requiring medical attention
Arm/Group | Treatment as Usual (TAU) + Internet | Treatment as Usual (TAU) + ElderTree
Number analyzed (Participants) | 168 | 176
falls requiring medical attention
  Baseline | 0.23 (0.50) | 0.18 (0.39)
  12-months | 0.33 (0.84) | 0.16 (0.37)

ADVERSE EVENTS:
Time Frame: up to 18 months
Arm/Group | Treatment as Usual (TAU) + Internet | Treatment as Usual (TAU) + ElderTree
All-Cause Mortality (participants affected / at risk) | 4/168 | 8/176
Serious Adverse Events (participants affected / at risk) | 0/168 | 0/176
Other Adverse Events (participants affected / at risk) | 0/168 | 0/176

LIMITATIONS AND CAVEATS:
We did not have health lab score baseline data for all participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT03387735/Prot_SAP_001.pdf
  • Informed Consent Form (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT03387735/ICF_000.pdf